CLINICAL TRIAL: NCT04130139
Title: Benefits of an Oocyte Pickup Simulation Training Program Using a High-fidelity Simulator for Obstetrics and Gynecology Residents
Brief Title: Benefits of an Oocyte Pickup Simulation Training Program
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pickupsim
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Simulation Training; IVf; Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- residents: obstetrics and gynecology residents from France with or without previous experience in oocyte pick up
  Interventions: Other: oocyte pick up simulator

INTERVENTIONS:
Other: oocyte pick up simulator — oocyte pick up simulation

SUMMARY:
The primary objective of this study was to evaluate oocyte pick up simulation training program for teaching residents. The secondary objectives were to evaluate resident satisfaction and the overall current state of oocyte pick up training in France.

DETAILED DESCRIPTION:
simulation workshop using PickupSim simulator. inclusion: obstetrics and gynecology residents from France simulator: 7 scenarios available

1 simulation training/resident main outcome: successful completion of the scenario (oocyte retrieval rate >=70%) secondary outcome: time for completion, complications, satisfaction survey

ELIGIBILITY:
Inclusion Criteria:

* obstetrics and gynecology residents
* french residents

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: obstetrics and gynecology residents from France participating in a national training conference organized by the national college of french gynecologists and obstetricians.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
successful scenario | 1 day
  oocyte retrieval rate >=70%

SECONDARY OUTCOMES:
completion time | 1 day
  time to successfully complete the scenario
complications | 1 day
  complications that may occurs during the simulation training (lesions of vitals organs, forget to change collection tubes)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Emmanuel Bouet, MD, Principal Investigator — Centre hospitalier d'Angers
Locations (1):
- Centre Hospitalier Universitaire Angers, Angers, France